CLINICAL TRIAL: NCT02115360
Title: The Pre-emptive Value of Epidural Calcitonin in Patients With Lower Limb Amputation. A Double Blinded Randomized Study
Brief Title: Epidural Calcitonin in Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2308/1/14
Record Dates: First submitted 2014-04-13; First posted 2014-04-16 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Amputation Stumps
Keywords: epidural calcitonin; amputation; postoperative pain; Later Complication
MeSH Terms: conditions — Pain, Postoperative | interventions — Calcitonin; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcitonin (Active Comparator): Under full aseptic conditions, the epidural space was identified at the L 2-3 or L 3-4 lumbar interspace using the loss-of-resistance to saline technique using 16-gauge Tuohy needle. A test-dose of 3 mL of a 2% solution of lidocaine with adrenaline (1:200,000) will be given to exclude subarachnoid or intravenous catheter placement. An injection of a2 ml hyperbaric bupivacaine will be injected into the subarachnoid space through 25 gauge spinal needle, then 15ml 0.5% bupivacaine, 100 micrograms of fentanyl and 100 iu of calcitonin will be injected epidurally in Bupivacain-Calcitonin-fentanyl (BC) Group,
  Interventions: Drug: Calcitonin
- fentanyl (Active Comparator): Under full aseptic conditions, the epidural space was identified at the L 2-3 or L 3-4 lumbar interspace using the loss-of-resistance to saline technique using 16-gauge Tuohy needle. A test-dose of 3 mL of a 2% solution of lidocaine with adrenaline (1:200,000) will be given to exclude subarachnoid or intravenous catheter placement. An injection of a2 ml hyperbaric bupivacaine will be injected into the subarachnoid space through 25 gauge spinal needle, then 15ml 0.5% bupivacaine, 100 micrograms of fentanyl and 1ml normal saline will be injected epidurally in Bupivacain- fentanyl (BF) Group, then a 16G Portex catheter was inserted for post- operative analgesia.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Calcitonin — Under full aseptic conditions, the epidural space was identified at the L 2-3 or L 3-4 lumbar interspace using the loss-of-resistance to saline technique using 16-gauge Tuohy needle. A test-dose of 3 mL of a 2% solution of lidocaine with adrenaline (1:200,000) will be given to exclude subarachnoid or intravenous catheter placement. An injection of a2 ml hyperbaric bupivacaine will be injected into the subarachnoid space through 25 gauge spinal needle, then 15ml 0.5% bupivacaine, 100 micrograms of fentanyl and 1ml normal saline will be injected epidurally in Bupivacain- fentanyl (BF) Group, then a 16G Portex catheter was inserted for post- operative analgesia.
  Other Names: maicalciac
  Arms: Calcitonin
Drug: Fentanyl — Under full aseptic conditions, the epidural space was identified at the L 2-3 or L 3-4 lumbar interspace using the loss-of-resistance to saline technique using 16-gauge Tuohy needle. A test-dose of 3 mL of a 2% solution of lidocaine with adrenaline (1:200,000) will be given to exclude subarachnoid or intravenous catheter placement. An injection of a2 ml hyperbaric bupivacaine will be injected into the subarachnoid space through 25 gauge spinal needle, then 15ml 0.5% bupivacaine, 100 micrograms of fentanyl and 1ml normal saline will be injected epidurally in Bupivacain- fentanyl (BF) Group, then a 16G Portex catheter was inserted for post- operative analgesia.
  Other Names: fentavera
  Arms: fentanyl

SUMMARY:
A prospective randomized double-blind clinical trial design will be used in a cohort of sixty patients of both genders, physical status American Society of Anaesthesiologist (ASA) I and II who will undergo lower limb amputation, will be enrolled into the present study. Patients will divided randomly into two equal groups: Epidural Bupivacain-Calcitonin and fentanyl (BC) Group and Bupivacain- fentanyl (BF) Group, comprising of 30 patients each.

DETAILED DESCRIPTION:
a cohort of sixty patients of both genders, physical status American Society of Anaesthesiologist (ASA) I and II who will undergo lower limb amputation, will be enrolled into the present study. Patients will divided randomly into two equal groups: Epidural Bupivacain-Calcitonin and fentanyl (BC) Group and Bupivacain- fentanyl (BF) Group, comprising of 30 patients each.

ELIGIBILITY:
Inclusion Criteria:

* prospective randomized double-blind clinical trial design will be used in a cohort of sixty patients of both genders
* physical status American Society of Anaesthesiologist (ASA) I and II
* will undergo lower limb amputation

Exclusion Criteria:

* history of pituitary gland dysfunction
* cardiac disease
* chronic obstructive respiratory disease
* contraindications to performing an epidural block such as:

  * coagulation abnormalities
  * spinal deformities, and
* patients allergic to local anesthetics and or calcitonin will be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 48 hours
  The primary outcome of the study the analgesic effects of epidural calcitonin versus opioids administered for patients undergoing lower limb amputation surgery on postoperative pain using combined spinal epidural anesthesia.

SECONDARY OUTCOMES:
Analgesic consumption | 48 hours
  The secondary outcome of this study is to measure analgesic consumption in patients undergoing lower limb amputation using combined spinal epidural anesthesia.

OTHER OUTCOMES:
post amputation pain | 6 months
  the development of post amputation phantom limb pain in calcitonin versus opioids administered for patients undergoing lower limb amputation surgery on postoperative pain using combined spinal epidural anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant Professor
Locations (1):
- Tanta University Hospitals, Tanta, Algharbyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Knopp-Sihota JA, Newburn-Cook CV, Homik J, Cummings GG, Voaklander D. Calcitonin for treating acute and chronic pain of recent and remote osteoporotic vertebral compression fractures: a systematic review and meta-analysis. Osteoporos Int. 2012 Jan;23(1):17-38. doi: 10.1007/s00198-011-1676-0. Epub 2011 Jun 10. PMID 21660557